CLINICAL TRIAL: NCT04915274
Title: Validation of an Electronic Remote Toxicity Management System in Adult Cancer Patients Receiving an Active Anti-cancer Treatment
Brief Title: Validation of an Electronic Remote Toxicity Management System in Cancer Patients
Acronym: eRToMSy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-01-CHRMT
Record Dates: First submitted 2021-05-17; First posted 2021-06-07 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Cancer
Keywords: Cancer; Active anticancer drug; Quality of life; QuestOnco application
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult cancer patients (Experimental): Patients will be provided with the QuestOnco application for monitoring
  Interventions: Other: uses of an application

INTERVENTIONS:
Other: uses of an application — Patients will be advised that they can still use their QuestOnco handset if they are hospitalized only for a treatment-related toxicity.

SUMMARY:
To assess the psychometric properties (validity, reliability and responsiveness) of the QuestOnco tool, an electronic Remote Toxicity Management System, in adult cancer patients receiving an active anti-cancer treatment.

DETAILED DESCRIPTION:
In this study, a mobile phone-based remote monitoring system (QuestOnco application) was developed in order to enable the 'real-time' monitoring of patients' symptoms through use of ePROMs. In order to establish if this new application accurately and reliably identifies the anti-cancer treatment related symptoms, its psychometric properties (validity, reliability and responsiveness) have to be assessed.

Hypotheses:

* The QuestOnco application will be designed as a promising innovative tool with good psychometric properties in order to detect more rapidly the anti-cancer-related toxicity in adult cancer patients.
* The QuestOnco application is an accurate and reliable tool for the identification of the anti-cancer treatment related symptoms as much as current available questionnaires such as PRO-CTCAE and EORTC QLC-QC30 The evaluation of the psychometric properties of the QuestOnco application will be made in two phases. First, the patient's cognitive interviews will allow assessing the content validity of the items. Then focus groups including patients and professional experts will determine the QuestOnco application goals regarding the adverse symptoms management (recommendations provided within the application, connection with General practitioner, medical Oncology team or Emergency departments).

This study will assess the validity, reliability and responsiveness of the QuestOnco in a cohort of patients receiving anti-cancer treatments. The external validity will be directly compared to PRO-CTCAE (Patient-Reported Outcome Common Terminology Criteria for Adverse Events) and to EORTC QLC-QC30 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years);
* Written and informed consent;
* Diagnosis of solid cancer;
* Metastatic or (neo)adjuvant anti-cancer treatment, including intravenous and/or oral treatments;
* Patient physically/psychologically fit to participate in the study;
* Patient able to understand, communicate and use the electronic device;
* Patient owning a smartphone or tablet with internet connection;
* Treatment supported by the French social security system.

Exclusion Criteria:

* Unable patient for signing informed consent;
* Unable to understand, communicate and use the electronic device;
* Patient under trusteeship or guardianship;
* Patient under legal or administration protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
Convergent validity | At the end of study completion (Week 6)
  PRO-CTCAE The convergent validity will be evaluated by the correlation between the QuestOnco and the weekly paper form of the PRO-CTCAE questionnaire.
  PRO-CTCAE is a patient-reported outcome (PRO) measurement system developed to evaluate symptomatic toxicity in patients on cancer clinical trials. It was designed to be used as a companion to the Common Terminology Criteria for Adverse Events (CTCAE) External Web Site Policy, the standard lexicon for adverse event reporting in cancer clinical trials.
  The PRO-CTCAE Item Library includes 124 items representing 78 symptomatic toxicities drawn from the CTCAE. PRO-CTCAE items evaluate the symptom attributes of frequency, severity, interference, amount, presence/absence. Each symptomatic AE is assessed by 1-3 attributes.
  PRO-CTCAE responses are scored from 0 to 4 (minimum/maximum).

SECONDARY OUTCOMES:
Patients' comprehension of QuestOnco application items | At the end of the study completion: Phase I (Day 7)
  Semi-structured cognitive interviews:
  Interviews will be conducted to evaluate patients' comprehension of the QuestOnco application items. Items will be modified and restested if more than 2 patients manifest cognitive difficulties. The item modifications will be conducted during focus groups gathering experts including Emergency department practitioners, General practitioner, Oncologists, Pharmacists, and Methodologists. This procedure will be repeated 3 times a maximum for a total of 30 patients.
The known-groups validity assessment | At the end of the study completion (Week 6)
  The known-groups validity will be assessed by comparing the QuestOnco items between patients with high and low performance status using the Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1 vs 2-4 (minimum vs maximum).
Evaluation of the efficacy of the QuestOnco application in patient care | At the end of study completion (Week 6)
  Calculation of the time spent (minutes) in consultation with the Oncologist using QuestOnco application fill form
Evaluation of the responsiveness of the QuestOnco application in patient care | At the end of the study completion (Week 6)
  Calculation of the number (percent) of appointments actually realized using QuestOnco application fill form
The reliability of the QuestOnco application in patient care | At the end of the study completion (Week 6)
  Calculation of the number (percent) of the automatic telephone alert calls to the regional Emergency service using QuestOnco application fill form
Synchronization of departments (Emergency division, Oncology team) and patients' care | At the end of the study completion (Week 6)
  Calculation of the number (percent) of scheduled consultation based on the statement of reported-toxicity score (symptom severity from grades II to IV) of cancer patients using electronic mobile QuestOnco application.
Evaluation of the Quality of Life of patients who use QuestOnco healthcare mobile application | At the end of the study completion (Week 1 and 6)
  The patients' quality of life will be assessed using EORTC QLC-QC30 questionnaire The EORTC QLQ-C30 is a 30-item core-cancer-specific questionnaire-integrating system for assessing the health-related QOL of cancer patients participating in international clinical trials. The questionnaire incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea and vomiting), a global health and QOL scale, and single items for the assessment of additional symptoms commonly reported by cancer patients (e.g., dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea), as well as the perceived financial impact of the disease and treatment. All items are scored on 4-point Likert scales, ranging from 1 ('not at all') to 4 ('very much'), with the exception of two items in the global health/QOL scale which use modified 7-point linear analog scales.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele LONGO, Principal Investigator — CHR METZ THIONVILLE; Véronique NOIREZ, Study Director — CHR METZ THIONVILLE
Locations (1):
- Centre Régional Metz-Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Longo R, Goetz C, Campitiello M, Plastino F, Egea J, Legros PO, Elnar AA, Meraihi S, Luporsi E, Noirez V. Content validation of an electronic remote toxicity management system in adult patients undergoing cancer treatment: a prospective longitudinal study on the QuestOnco application. BMC Cancer. 2024 Dec 23;24(1):1568. doi: 10.1186/s12885-024-13312-4. PMID 39716103